CLINICAL TRIAL: NCT01303562
Title: Clinical Assessment of Barley and Oat Phytochemicals: Acute Bioavailability, Pharmacokinetics, and Bioactivity
Brief Title: Clinical Assessment of Barley and Oat Phytochemicals
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tufts University (Other)
Collaborators: Kellogg Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: IRB 9571
Record Dates: First submitted 2010-11-16; First posted 2011-02-24 (Estimated); Last update posted 2013-05-27 (Estimated); Status verified 2013-05

CONDITIONS: Healthy
Keywords: oat; barley; whole grain; bioavailability; phytochemical
MeSH Terms: conditions — Gyrate Atrophy

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (3):
- Placebo muffin made with no whole grains (Placebo Comparator)
  Interventions: Other: Whole grain oats and barley
- Test muffin made with whole oats (Active Comparator)
  Interventions: Other: Whole grain oats and barley
- Test muffin made with whole barley (Active Comparator)
  Interventions: Other: Whole grain oats and barley

INTERVENTIONS:
Other: Whole grain oats and barley — One time dose of 48 g whole grain flour in 2 small muffins (24 g flour per muffin) per intervention

SUMMARY:
The goal of this placebo-controlled, 3-way crossover study is to determine the acute (24-h) bioavailability and pharmacokinetics of the major phytochemicals found whole barley and oats, as well as their effects on selected measures of antioxidation, inflammation, insulin sensitivity/glucose regulation, and vascular remodeling following challenge by an oral glucose tolerance test (OGTT).

ELIGIBILITY:
Inclusion Criteria:

* Men and postmenopausal women
* BMI 27-35.9 kg/m2

Exclusion Criteria:

* Cigarette smoking and/or nicotine replacement use
* Individuals taking estrogen
* Use of cholesterol-lowering medications
* Use of blood pressure-lowering medications
* Regular use of any stomach acid-lowering medications or laxatives (including fiber supplements)
* Cardiovascular (heart) disease
* Gastrointestinal disease
* Kidney disease
* Endocrine disease: including diabetes, untreated thyroid disease
* Rheumatoid arthritis
* Active treatment for any type of cancer, except basal cell carcinoma, within 1 year prior to study admission
* Systolic blood pressure > 150 mmHg and/or diastolic blood pressure > 95 mmHg
* Regular use of oral steroids
* Regular daily intake of ≥ 2 alcoholic drinks
* Infrequent or excessive number of regular bowel movements
* Illicit drug use
* Vegetarians
* No fish oil supplements (including cod liver oil) for one month prior to study admission
* No dietary supplements, including those containing any vitamins, minerals, herbs, plant concentrates (including garlic, gingko, St. John's wort) or homeopathic remedies, for one month prior to study admission

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2010-09; Primary Completion 2011-04 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Levels of phytochemicals and their in vivo metabolites in blood | 24 hours
  Levels of phytochemicals and their in vivo metabolites in blood, urine, and feces following the consumption of whole grains delivered in a baked muffin

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey B Blumberg, PhD, Principal Investigator — Tufts Medical Center
Locations (1):
- Tufts Clinical and Translational Research Center, Boston, Massachusetts, United States